CLINICAL TRIAL: NCT03684720
Title: Using 'Guided-Discovery-Learning' to Optimize and Maximize Transfer of Surgical Simulation
Acronym: GDLEFFICACY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Andreas Höier Aagesen, Principle Investigator, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GDL-Efficacy
Record Dates: First submitted 2018-08-24; First posted 2018-09-26 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Humans; Simulation Training; Problem-Based Learning; Clinical Competence; Education, Medical; Learning; Surgical Procedure, Unspecified
Keywords: Medical education; Basic Science; Procedural skills; Simulation; Transfer; Instructional design; Guided Discovery Learning; Retention

STUDY DESIGN:
Intervention Model Description: The study is a randomized experimental study comparing 2 groups, a control and an intervention. One group will receive traditional instructional teaching (control) and the other will receive guided-discovery-learning (intervention). Both groups will undertake the same tests after the teaching session.
Who Masked: Outcomes Assessor
Masking Description: The groups will be masked, until the day of the teaching session, so the investigator won't know, which group he assigns participants to, when enrolling them. The raters who will score the participants, will have no knowledge of which group the participant belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discover followed by direct instruction [DD] (Experimental): The intervention group which will be taught suturing using guided-discovery-learning
  Interventions: Other: Discover followed by direct instruction [DD]
- Instruction followed by practice [IP] (No Intervention): The control group which will be taught suturing using traditional instructional teaching.

INTERVENTIONS:
Other: Discover followed by direct instruction [DD] — The intervention group will be taught suturing using the principles of guided-discovery-learning. In its simplest form, this means allowing the participants to practice placing a simple interrupted suture using the materials needed, as well as a picture of a finished suture. They must then draw from their own learning experiences, as well as discover for themselves how to do it. After a discovery period, an instructor will then teach them, how to place a simple interrupted suture, and will them guide them, as they begin to practice again.
  Other Names: Guided-discovery-learning
  Arms: Discover followed by direct instruction [DD]

SUMMARY:
The study is a randomized experimental study comparing two forms of learning; guided-discovery-learning and traditional instructional learning. Recruiting sixty-four participants, the investigators plan on comparing these two groups through a procedural skill in the form of suturing. In the case of guided-discovery-learning, the group will be allowed a discovery phase before instruction. In contrast, the control group will receive traditional instruction-lead-learning, in which a teacher teaches the participants a skill, and afterwards the participants practice it. After the teaching session, both groups will undertake a post-test of skill-level. A week later both groups will undertake a test for the execution of the learned suturing skill to a more complex version of the original task (Near-transfer). They will also undergo a test for the ability to transfer their learning to a new skill (i.e. preparation for future learning), in this case a new suture (Far-transfer). By filming these tests and having a blinded expert rater score them, the investigators will be able to get a measurement of attained transfer of skill-level throughout the procedures. The investigators hypothesis is that, the participants in the Guided-discovery-group will have an equal score to that of the traditional-learning group in the ability to obtain a skill and transfer it to a more complex version. Furthermore, the investigators hypothesize that the Guided-discovery-group will score better than the traditional-learning group in the case of transferring the procedural knowledge to learning a new skill.

As well as testing the efficacy of guided-discovery-learning on a procedural skill, the investigators wish to investigate how and why it works. By filming a subset of participants in each group, as well as using questionnaires, and focus-group interviews the investigators will explore how participants interact in this different learning-environment compared to the traditional instructional learning-environment.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Technical skills are a core competency in surgical specialties. The level of technical skills is directly linked to patient outcomes and it is an absolute requirement that surgical trainees learn to master basic surgical skills. It is therefore a necessity that medical students also become well equipped with these skills, such as suturing. During the last decade, minimally invasive techniques have made their way to the operating room and improved patient outcomes. Despite these advances it is still necessary for surgeons to master the open surgical skills. Unexpected complication can arise in minimally invasive procedures that require conversion to open access surgery. Furthermore, there are procedures where you cannot use minimally invasive techniques. Because of the extensive use of minimally invasive surgery, it is becoming more difficult for doctors as well as medical students in surgical departments to gain the level of experience needed, to become proficient in open surgical techniques. Pre-clinical teaching and simulation training is a possible solution to this problem For novice learners, simulation training is an opportunity to acquire fundamental skills such as suturing in a safe and high-feedback environment and without the difficulties of acquiring these skills in the workplace. For more advanced trainees, simulation affords the practice of difficult and complex procedures which may be otherwise too unsafe to acquire during patient care. But, merely implementing simulation training is no guarantee of educational utility, and instead thoughtful curricular integration of simulation requires considering the role and purpose of the simulator, the student experience, debriefing, and the intended outcomes to evaluate success.

One potential area for optimizing simulation-based training is to clarify instructors' roles when providing guidance and direct supervision. One of the challenges with simulation training is the amount of resources this sort of education requires. Especially the amount of time a student spends interacting with an instructor. Supervision and instruction are key to an effective simulation-based training, and there is mounting evidence, which suggest, that the community needs to reconsider the balance between instruction and discovery, allowing for a good interaction between student and teacher, encouraging learning. Therefore the question is; on what level should simulation-based teaching be instructor-orientated? When teaching technical medical skills, the answer to the question, whether the training should be discovery-orientated or instructor-orientated has been thoroughly researched. Medical Education literature has long moved away from the question of either or, and is now more focused on, in which order discovery- and instruction-teaching should be, to provide the best learning outcome. Recent studies has shown some positive results of guided-discovery-learning, which in its simple form, combines both elements from discovery and instruction-based teaching. Especially the ability to 'transfer' learning seems vastly improved, with this teaching method. Transfer tasks faced by learners exist on spectrum with a common challenge being new problems which are more complex or in new contexts but essentially require replication of previously learned skills, i.e. near transfer. While near transfer can be difficult for learners, even more challenging is transfer that requires they apply their previous skills and understanding to learn new skills or concepts, i.e. far transfer. Guided-discovery learning has been shown to especially positively impact this latter type of transfer task. Thus guided-discovery may promote student-autonomy and self-learning which subsequently enables students to take responsibility for their own future learning.

In a pilot-study completed by the investigators research-partners at the Wilson-Centre in Toronto, Canada, they compared groups of discovery followed by direct discovery (DD) with instruction followed by discovery (IP). In the case of DD, the participants, where given the materials needed to complete a simple suture, and a finished suture to look at. After the discovery-phase, they were parred with an instructor who demonstrated how it was to be performed. In the IP-case they were first instructed on how to perform the suture, and were afterwards allowed to practice it. At the end of the course both groups were given a post-test of ability, and a week-later both groups were given a retention test as well as a transfer test. The pilot-study included 26 participants in total, divided in two groups of 13. The participants were randomized, and everything was filmed and scored by blinded raters after an international standard. There were no significant results for the immediate post-test as well as the retention test. But in the case of the transfer test, the DD-group was far superior.

The investigators study will expand on the pilot-study to provide a comparison of guided discovery to traditional instruction for the learning of suturing tasks in surgery, seeing if Guided-discovery-learning works in a much larger research group. Using a double randomized, mixed-methods experimental design, the investigators will investigate the effect of discovery followed by direct instruction (DD) vs. instruction followed by practice (IP) for the acquisition and two types of transfer of surgical skills.

The investigators hypothesize that:

1. Participants in the DD condition will be better able to transfer their knowledge to learning a new skill (i.e., preparation for future learning).
2. Participants in the DD condition will have equivalent performance to IP on post-test, but a similar or slightly improved performance on transfer of suturing skill to a more complex task (near-transfer).
3. Participants in the DD condition will interact differently with instructors and will use their learnings from the discovery phase to scaffold their learning during the direct instruction phase as well as interacting differently with the task at hand.

EXPERIMENTAL DESIGN:

The study will be performed at CAMES, including n=64 pre-clinical medical students from the Copenhagen University. The investigators are targeting undergraduate students, rather than surgical residents, because they want novice learners, and they believe it is worthwhile to establish efficacy of the intervention group using simpler tasks which can be feasibly studied. The investigators based their sample size on the previous pilot-study which suggests that detecting a large effect on a global rating scale (Hedges g of >0. with an alpha of 0.05 and power of 80% requires at least 13 participants per group with additional participants recruited for potential loss to follow-up for a total of 16 per group. Participants will receive a certificate showing completed suturing course, as an honorarium to compensate for their time in the study.

Part 1 of this study is an experimental design with two phases that will test the efficacy of guided discovery: Phase 1 will be a learning phase with the experimental manipulations, and Phase 2 will take place one week later and be outcome assessment for near- and far transfer. Part 2 of this study will be explorative seeking answers to how and why guided-discovery works.

For Phase 1, participants will be enrolled and randomly allocated to either the DD or IP groups. Each group consists of 8 participants. Participants will be randomized and the method of teaching allocated on the date of teaching. This will ensure generalization and ease of statistical analysis. In the DD group, participants will be given an example of a completed simple interrupted suture and their own skin pad, and suturing kit. They will then attempt to replicate the suture using the equipment and their own knowledge over 30 minutes. During the same period of time, the IP group will be taught using an instructor. The instructor will provide two demonstrations and explanations of the simple interrupted suture following which the participants will attempt the suture individually on their own skin pads and suturing kit (Modifications will be made by an experienced surgical instructor on our team ST). The instructor will be told to provide feedback and guidance to the participants as well as answer any questions that participants may have. After the initial time, the DD group will be paired with an instructor who will provide two demonstrations and explanations of the suture and then interact with participants as they attempt the suture. The IP group will practice the suture without any further instructor guidance. At the end of the teaching session, all participants will complete a post-test requiring them to complete two simple interrupted sutures. Afterwards participants willing will be interview in short focus-group interviews. This entire session is expected to last 2 hours including consent and setup time.

After a 1-week delay, participants will return for Phase 2 for the tests of near- and far transfer. Each group will again be randomly allocated a transfer task. Two transfer tasks will be used in this study: To test Hypothesis 1, (the impact on transfer to future learning), participants will be taught the interrupted vertical mattress suture. To ensure equivalency of design and to prevent biasing in favor of one group, all participants will be taught didactically, which will involve viewing a 15-minute video designed by an expert surgeon on our team (ST) to teach the novel suturing task. Participants will then be given 20-30 minutes to practice the suture following which they will perform two vertical matrass sutures on a typical skin pad.

To test Hypothesis 2 (the impact on transfer of learning to a more complex version of the initial task) participants will perform two simple interrupted sutures on a suturing pad representing in an abdominal simulator with the added contextual change of different instruments and suture. In both groups, participants willing, will afterwards be recorded for a 'Think-Aloud' interview, in which they describe their approach to the suturing task out-loud. This phase is expected to last 1.5 hours.

PERSPECTIVES:

Faculty instructors are a limited resource in formal simulation-based training during post-graduate training. The rise of structured learning activities such as surgical boot camps and the emphasis on greater feedback and support for trainees means that instructor time is at a greater premium than ever before. Instructors must take time away from their busy clinical and workplace-based education activities in order to teach. Not only does this cost the healthcare system, the time commitment can reduce willingness to participate in education. Additional costs may be incurred by programs that must offer financial incentives for instructors. This trade-off between education and clinical work occurs in all academic postgraduate programs. Given the cost and investment required to recruit faculty for training, research is needed to maximize the efficiency of faculty involvement. The investigators work directly contributes to this goal by identifying how instructor guidance is most helpful to trainees. Guided-discovery may be one approach to reducing the cost of training and instructor time in both post-graduate as well as pre-graduate learning courses.

Post-graduate training also requires that trainees develop autonomy and are able to learn new skills or concepts effectively (stresses trainees' abilities to transfer their training when faced with uncertainty and or complexity in future scenarios. Guided-discovery may be an effective organizing principle for educational design that can achieve these competencies across a wide range of disciplines and training environments. The investigators proposal would thus establish evidence of efficacy for guided-discovery for these competency roles.

ELIGIBILITY:
Inclusion Criteria:

* Participant are students currently attending a Danish medical bachelor and who are willing and consent to participation in the study.

Exclusion Criteria:

* Participants who have received prior suturing education are excluded from participating in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Effects of Guided-Discovery-Learning in the Far Transfer of Simple Surgical Skills. | Through study completion on average 12 months
  Comparison of far transfer-test between control and intervention group as assessed by OSATS: Global Rating Scale of Performance. OSATS is short for: Objective Structured Assessment of Technical Skills. It consists of 7 subsets of which 5 are relevant to the study. Each participant is rated from 1(minimum) to 5(maximum) in each subset, and all subsets are added together by simple summation. This gives the participants a total score of out of 25 points, where the higher the number the better the performance.

SECONDARY OUTCOMES:
Effects of Guided-Discovery-Learning on the Near Transfer of Simple Surgical Skills. | Through study completion on average 12 months
  Comparison of near transfer-test between control and intervention group as assessed by OSATS: Global Rating Scale of Performance. OSATS is short for: Objective Structured Assessment of Technical Skills. It consists of 7 subsets of which 5 are relevant to the study. Each participant is rated from 1(minimum) to 5(maximum) in each subset, and all subsets are added together by simple summation. This gives the participants a total score of out of 25 points, where the higher the number the better the performance.
Effects of Guided-Discovery-Learning immediately after a training-session in simple surgical skills. | Through study completion on average 12 months
  Comparison of post-test skill level between control and intervention group as assessed by OSATS: Global Rating Scale of Performance. OSATS is short for: Objective Structured Assessment of Technical Skills. It consists of 7 subsets of which 5 are relevant to the study. Each participant is rated from 1(minimum) to 5(maximum) in each subset, and all subsets are added together by simple summation. This gives the participants a total score of out of 25 points, where the higher the number the better the performance.
Impact Difference on near and far transfer using Guided-Discovery-Learning | Through study completion on average 10 months
  Comparison of near and far transfer scores in both control and intervention groups [change from baseline post-test to near- and far transfer tests] using OSATS: Global Rating Scale of Performance. OSATS is short for: Objective Structured Assessment of Technical Skills. It consists of 7 subsets of which 5 are relevant to the study. Each participant is rated from 1(minimum) to 5(maximum) in each subset, and all subsets are added together by simple summation. This gives the participants a total score of out of 25 points, where the higher the number the better the performance.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas H Aagesen, Principal Investigator — Copenhagen Academy for Medical Education and Simulation
Locations (1):
- Copenhagen Academy of Medical Education and Simulation, Copenhagen, KBH Ø, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reznick RK, MacRae H. Teaching surgical skills--changes in the wind. N Engl J Med. 2006 Dec 21;355(25):2664-9. doi: 10.1056/NEJMra054785. No abstract available. PMID 17182991
- [Background] Dawe SR, Pena GN, Windsor JA, Broeders JA, Cregan PC, Hewett PJ, Maddern GJ. Systematic review of skills transfer after surgical simulation-based training. Br J Surg. 2014 Aug;101(9):1063-76. doi: 10.1002/bjs.9482. Epub 2014 May 15. PMID 24827930
- [Background] Zendejas B, Brydges R, Hamstra SJ, Cook DA. State of the evidence on simulation-based training for laparoscopic surgery: a systematic review. Ann Surg. 2013 Apr;257(4):586-93. doi: 10.1097/SLA.0b013e318288c40b. PMID 23407298
- [Background] Zendejas B, Cook DA. Reply to Letter: "Surgical Simulation: Seeing the Bigger Picture and Asking the Right Questions". Ann Surg. 2015 Aug;262(2):e51-2. doi: 10.1097/SLA.0000000000001138. No abstract available. PMID 25607763
- [Background] Brydges R, Nair P, Ma I, Shanks D, Hatala R. Directed self-regulated learning versus instructor-regulated learning in simulation training. Med Educ. 2012 Jul;46(7):648-56. doi: 10.1111/j.1365-2923.2012.04268.x. PMID 22691145
- [Background] Brydges R, Dubrowski A, Regehr G. A new concept of unsupervised learning: directed self-guided learning in the health professions. Acad Med. 2010 Oct;85(10 Suppl):S49-55. doi: 10.1097/ACM.0b013e3181ed4c96. PMID 20881703
- [Background] Lee HS, Anderson JR. Student learning: what has instruction got to do with it? Annu Rev Psychol. 2013;64:445-69. doi: 10.1146/annurev-psych-113011-143833. Epub 2012 Jul 12. PMID 22804771
- [Background] Mylopoulos M, Brydges R, Woods NN, Manzone J, Schwartz DL. Preparation for future learning: a missing competency in health professions education? Med Educ. 2016 Jan;50(1):115-23. doi: 10.1111/medu.12893. PMID 26695471
- [Background] DeCaro MS, Rittle-Johnson B. Exploring mathematics problems prepares children to learn from instruction. J Exp Child Psychol. 2012 Dec;113(4):552-68. doi: 10.1016/j.jecp.2012.06.009. Epub 2012 Jul 31. PMID 22849809
- [Background] Grierson LE. Information processing, specificity of practice, and the transfer of learning: considerations for reconsidering fidelity. Adv Health Sci Educ Theory Pract. 2014 May;19(2):281-9. doi: 10.1007/s10459-014-9504-x. Epub 2014 Apr 2. PMID 24691891
- [Background] Hatala R, Cook DA, Brydges R, Hawkins R. Constructing a validity argument for the Objective Structured Assessment of Technical Skills (OSATS): a systematic review of validity evidence. Adv Health Sci Educ Theory Pract. 2015 Dec;20(5):1149-75. doi: 10.1007/s10459-015-9593-1. Epub 2015 Feb 22. PMID 25702196
- [Background] Devine LA, Donkers J, Brydges R, Perelman V, Cavalcanti RB, Issenberg SB. An Equivalence Trial Comparing Instructor-Regulated With Directed Self-Regulated Mastery Learning of Advanced Cardiac Life Support Skills. Simul Healthc. 2015 Aug;10(4):202-9. doi: 10.1097/SIH.0000000000000095. PMID 26154249
- [Background] Brydges R, Manzone J, Shanks D, Hatala R, Hamstra SJ, Zendejas B, Cook DA. Self-regulated learning in simulation-based training: a systematic review and meta-analysis. Med Educ. 2015 Apr;49(4):368-78. doi: 10.1111/medu.12649. PMID 25800297

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT03684720/Prot_SAP_ICF_002.pdf